CLINICAL TRIAL: NCT05423730
Title: Effect of Light Alcohol Intake on Sex Hormone Levels Among Postmenopausal Women With ER+ Breast Cancer on Aromatase Inhibitor Therapy: The Alcohol and Breast Cancer (ABC) Trial
Brief Title: Alcohol and Breast Cancer (ABC) Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Kenneth Mukamal, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 21-698; K01AA027831 (NIH)
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: ER+ Breast Cancer; Breast Cancer; Aromatase Inhibitors
Keywords: ER+ Breast Cancer; Breast Cancer; Aromatase Inhibitors; Anastrozole; Letrozole; Exemestane
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WHITE WINE FOLLOWED BY WHITE GRAPE JUICE (Experimental): Participants will be randomized into one of the study drinking sequence groups: white wine followed by white grape juice or white grape juice followed by white wine.
  The research study procedures include one screening visit to obtain informed consent, four study visits with blood draws, and ten weekly phone calls and online questionnaires over the ten weeks of the study.
  -3 weeks of daily white wine followed by 3 weeks of daily white grape juice
  Interventions: Other: White Wine; Other: Grape Juice
- WHITE GRAPE JUICE FOLLOWED BY WHITE WINE (Experimental): Participants will be randomized into one of the study drinking sequence groups: white grape juice followed by white wine.
  The research study procedures include one screening visit to obtain informed consent, four study visits with blood draws, and ten weekly phone calls and online questionnaires over the ten weeks of the study.
  - 3 weeks of daily white grape juice followed by 3 weeks of daily white wine
  Interventions: Other: White Wine; Other: Grape Juice

INTERVENTIONS:
Other: White Wine — One serving (5 ounces) of white wine daily for 3 weeks
Other: Grape Juice — One serving (6 ounces) of white grape juice daily for 3 weeks

SUMMARY:
This research study is a pilot study, which is the first time investigators are examining the effect of light alcohol consumption on sex hormones among postmenopausal women with estrogen receptor-positive (ER+) breast cancer taking an aromatase inhibitor

The names of the study exposures involved in this study are:

* White wine
* White grape juice

DETAILED DESCRIPTION:
This research study is trying to to help understand whether light alcohol consumption causes short-term changes in the levels of estrogen, progesterone and testosterone, called sex hormones, among postmenopausal women with estrogen and/or progesterone receptor positive breast cancer taking estrogen-blocking medications called aromatase inhibitors.

The research study procedures include one screening visit to obtain informed consent, four study visits with blood draws, and ten weekly phone calls and online questionnaires over the ten weeks of the study.

This research study involves 10 weeks of participation, including 3 weeks consuming one serving of white wine daily, 3 weeks consuming one serving of white grape juice daily, and 2 weeks of drinking neither alcohol nor grape juice before each of these 3-week drinking periods.

In this experimental study, participants will be asked to drink white wine and white grape juice, which are not consumed as the standard of care. The U.S. Food and Drug Administration (FDA) has not approved alcohol as a treatment for any disease.

It is expected that about 20 women will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* ER+ breast cancer
* Female sex at birth
* Postmenopausal, either natural or induced
* Self-reported consumption of at least one alcoholic drink per week but not more than one serving per day
* Currently prescribed aromatase inhibitors including anastrozole (Arimidex®), letrozole (Femara®), and exemestane (Aromasin®)
* Documented liver function test results below 1.5X the upper limit of normal within 12 months of screening

Exclusion Criteria:

* Self-reported consumption of more than one drink per day, a previous or current history of alcohol abuse based on standard questionnaires (AUDIT≥8), or consumption of more than 4 or more drinks in one day within the last 6 months
* Currently undergoing cytotoxic chemotherapy or radiation or planned in the next two months
* Any surgery planned in the next two months
* Alcohol flushing syndrome
* Current use of any pharmaceutical agent contraindicated with alcohol, including warfarin, dual antiplatelet therapy, and metronidazole
* Hemoglobin A1c>8% or a fasting glucose result above 180 mg/dL within 6 months of screening
* Unable to speak or understand English
* Unable to understand and provide informed consent, as judged by the study team

Ages: 21 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Mukamal, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu

REFERENCES:
- [Derived] Mostofsky E, Buring JE, Come SE, Tung NM, Zhang C, Mukamal KJ. Effect of daily alcohol intake on sex hormone levels among postmenopausal breast cancer survivors on aromatase inhibitor therapy: a randomized controlled crossover pilot study. Breast Cancer Res. 2025 Jan 9;27(1):5. doi: 10.1186/s13058-024-01940-4. PMID 39789640

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We sent invitation letters to women taking AIs who received outpatient care at Beth Israel Deaconess Medical Center. Participants completed the study between September 2022 and July 2023.
Pre-assignment Details: Twenty-three participants consented to participate. Two participants drank too much to be eligible for the trial, and one declined to participate. All twenty women who were randomized completed the trial and are included in the analyses.
Groups:
- WHITE WINE FOLLOWED BY WHITE GRAPE JUICE: Participants will be randomized into one of the study drinking sequence groups: white wine followed by white grape juice or white grape juice followed by white wine.
  The research study procedures include one screening visit to obtain informed consent, four study visits with blood draws, and ten weekly phone calls and online questionnaires over the ten weeks of the study.
  -3 weeks of daily white wine followed by 3 weeks of daily white grape juice
  White Wine: One serving (5 ounces) of white wine daily for 3 weeks
  Grape Juice: One serving (6 ounces) of white grape juice daily for 3 weeks
- WHITE GRAPE JUICE FOLLOWED BY WHITE WINE: Participants will be randomized into one of the study drinking sequence groups: white grape juice followed by white wine.
  The research study procedures include one screening visit to obtain informed consent, four study visits with blood draws, and ten weekly phone calls and online questionnaires over the ten weeks of the study.
  - 3 weeks of daily white grape juice followed by 3 weeks of daily white wine
  White Wine: One serving (5 ounces) of white wine daily for 3 weeks
  Grape Juice: One serving (6 ounces) of white grape juice daily for 3 weeks
Period: Overall Study
Arm/Group | WHITE WINE FOLLOWED BY WHITE GRAPE JUICE | WHITE GRAPE JUICE FOLLOWED BY WHITE WINE
Started | 9 | 11
Completed | 9 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Crossover of White Wine and White Grape Juice: Participants will be randomized into one of the study drinking sequence groups: white wine followed by white grape juice or white grape juice followed by white wine.
  The research study procedures include one screening visit to obtain informed consent, four study visits with blood draws, and ten weekly phone calls and online questionnaires over the ten weeks of the study.
  -3 weeks of daily white wine followed by 3 weeks of daily white grape juice
  White Wine: One serving (5 ounces) of white wine daily for 3 weeks
  Grape Juice: One serving (6 ounces) of white grape juice daily for 3 weeks
Arm/Group | Crossover of White Wine and White Grape Juice
Number analyzed (Participants) | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61.0 [50 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
Total Estradiol Concentration [Median (Inter-Quartile Range); unit: pg/mL] | 0.8 [0.3 to 1.4]
Free Estradiol Concentration [Median (Inter-Quartile Range); unit: pg/mL] | 0.014 [0.005 to 0.02]
Free Estradiol Index [Median (Inter-Quartile Range); unit: pg/mL] | 0.012 [0.005 to 0.04]
Estrone [Median (Inter-Quartile Range); unit: pg/mL] | 0.9 [0.7 to 2.1]
Dehydroepiandrosterone Sulfate (DHEAS) [Median (Inter-Quartile Range); unit: ug/dL] | 57.5 [35.9 to 101.8]
Testosterone [Median (Inter-Quartile Range); unit: ng/dL] | 15.3 [11.7 to 25.2]
Sex hormone-binding globulin (SHBG) [Median (Inter-Quartile Range); unit: nmol/L] | 56.8 [29.7 to 92.1]

OUTCOME MEASURES:

1. Primary Outcome: Blood Levels of Total Estradiol Concentration
Description: Blood levels were measured at the beginning and end of three weeks of one serving (5 ounces) of white wine daily and the beginning and end of three weeks of one serving of white grape juice (6 oz) daily, with a two-week washout period before each drinking period. Estimates for levels following three weeks adjusted for blood levels at the beginning of the drinking period.
Time Frame: 3 Weeks
Population: We imputed values for estradiol below the lower limit of detection (0.5 pg/mL ) at one-half of that value. No other hormones fell below that value.
Measure: Least Squares Mean (95% Confidence Interval); unit: Log scale, pg/mL
Groups:
- White Grape Juice: One serving (6 ounces) of white grape juice daily for 3 weeks
Arm/Group | White Wine | White Grape Juice
Number analyzed (Participants) | 20 | 20
Log scale, pg/mL | -0.50 [-1.03 to 0.02] | -0.39 [-.91 to 0.14]
Statistical Analysis 1: Comparison: White Wine vs White Grape Juice; Test type: Superiority; Mean Difference (Final Values) = -11.12, 95% CI 2-sided [-49.75 to 57.20] — Estimates represent percentage change in log-transformed hormone levels for wine versus grape juice from linear mixed models including participant as a random effect and interaction terms for drink and sequence (Kenward approach)

2. Secondary Outcome: Blood Levels of Free Estradiol Concentration
Description: Blood levels were measured at the beginning and end of three weeks of one serving (5 ounces) of white wine daily and the beginning and end of three weeks of one serving of white grape juice (6 oz) daily, with a two-week washout period before each drinking period. Estimates for levels following three weeks adjusted for blood levels at the beginning of the drinking period. Estimates of free estradiol concentration were calculated using Mazer transformation.
Time Frame: 3 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Log scale, pg/mL
Arm/Group | White Wine | White Grape Juice
Number analyzed (Participants) | 20 | 20
Log scale, pg/mL | -4.53 [-5.10 to -3.96] | -4.45 [-5.03 to -3.88]
Statistical Analysis 1: Comparison: White Wine vs White Grape Juice; Test type: Superiority; Mean Difference (Final Values) = 7.65, 95% CI 2-sided [-47.96 to 63.90] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Blood Levels of Free Estradiol Index
Description: Estimated as total estradiol concentration divided by SHBG levels.Blood levels were measured at the beginning and end of three weeks of one serving (5 ounces) of white wine daily and the beginning and end of three weeks of one serving of white grape juice (6 oz) daily, with a two-week washout period before each drinking period. Estimates for levels following three weeks adjusted for blood levels at the beginning of the drinking period.
Time Frame: 3 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Log scale, pg/mL
Arm/Group | White Wine | White Grape Juice
Number analyzed (Participants) | 20 | 20
Log scale, pg/mL | -0.01 [-0.03 to 0.01] | 0 [-0.03 to 0.02]
Statistical Analysis 1: Comparison: White Wine vs White Grape Juice; Test type: Superiority; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-1.95 to 0.67] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Blood Levels of Estrone Concentration
Description: as for outcome 1
Time Frame: 3 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Log scale, pg/mL
Arm/Group | White Wine | White Grape Juice
Number analyzed (Participants) | 20 | 20
Log scale, pg/mL | 0.03 [-0.33 to 0.39] | -0.10 [-0.45 to 0.26]
Statistical Analysis 1: Comparison: White Wine vs White Grape Juice; Test type: Superiority; Mean Difference (Final Values) = 13.83, 95% CI 2-sided [-9.45 to 43.09] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Blood Levels of Dehydroepiandrosterone Sulfate (DHEAS)
Description: as for outcome 1
Time Frame: 3 Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Log scale, ug/dL
Arm/Group | White Wine | White Grape Juice
Number analyzed (Participants) | 20 | 20
Log scale, ug/dL | 4.18 [3.88 to 4.49] | 4.08 [3.77 to 4.38]
Statistical Analysis 1: Comparison: White Wine vs White Grape Juice; Test type: Superiority; Mean Difference (Final Values) = 11.42, 95% CI 2-sided [-3.31 to 28.40] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Blood Levels of Testosterone
Description: as for outcome 1
Time Frame: 3 Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Log scale, ng/dL
Arm/Group | White Wine | White Grape Juice
Number analyzed (Participants) | 20 | 20
Log scale, ng/dL | 2.75 [2.30 to 3.20] | 2.63 [2.18 to 3.09]
Statistical Analysis 1: Comparison: White Wine vs White Grape Juice; Test type: Superiority; Mean Difference (Final Values) = 12.57, 95% CI 2-sided [-0.77 to 27.69] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Blood Levels of Sex Hormone Binding Globulin (SHBG)
Description: as for outcome 1
Time Frame: 3 Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Log scale, nmol/L
Arm/Group | White Wine | White Grape Juice
Number analyzed (Participants) | 20 | 20
Log scale, nmol/L | 3.87 [3.49 to 4.26] | 3.90 [3.51 to 4.28]
Statistical Analysis 1: Comparison: White Wine vs White Grape Juice; Test type: Superiority; Mean Difference (Final Values) = -2.70, 95% CI 2-sided [-21.92 to 21.24] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | White Wine | White Grape Juice
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
This was a pilot trial with a small sample size and short treatment and washout periods.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-01-19): https://cdn.clinicaltrials.gov/large-docs/30/NCT05423730/Prot_SAP_ICF_000.pdf